CLINICAL TRIAL: NCT06437639
Title: Prospective, Open, Comparative, Randomized Study of the Efficacy and Safety Evaluation of the Mexidol® Sequential Therapy of Patients With Primary Open-angle Glaucoma (POAG)
Brief Title: MEXIDOL® Sequential Therapy of Patients With Primary Open-angle Glaucoma (POAG)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pharmasoft (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MexidolPOAG2024
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Primary Open-Angle Glaucoma (POAG)
Keywords: Glaucoma; Primary Open-Angle Glaucoma (POAG); Glaucomatous Optic Neuropathy (GON); Mitochondrial Dysfunction; Neuroprotection; Mexidol; Ethylmethylhydroxypyridine Succinate
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma; Mitochondrial Diseases | interventions — emoxypine succinate; ethylmethylhydroxypyridine succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Main (Mexidol and standard therapy) (Active Comparator): Mexidol IM 300 mg for 14 days, then Mexidol FORTE 250 orally 250 mg 1 tablet 3 times a day for 8 weeks; IOP normalizing therapy
  Interventions: Drug: Mexidol
- Control (standard therapy) (No Intervention): IOP normalizing therapy

INTERVENTIONS:
Drug: Mexidol — Neurocytoprotector
  Other Names: Ethylmethylhydroxypyridine Succinate
  Arms: Main (Mexidol and standard therapy)

SUMMARY:
Hypothesis: The use of neurocytoprotectors helps restore the functional activity of mitochondria, improve the nervous activity of the retina and optic nerve, and stabilize the glaucomatous process.

DETAILED DESCRIPTION:
Hypothesis: Mexidol® allows to optimize POAG therapy by reducing mitochondrial dysfunction and stabilizing glaucomatous optic neuropathy by improving the functional activity of mitochondria and its energy-producing function

ELIGIBILITY:
Inclusion Criteria:

* An advanced stage of POAG in one or two eyes
* Hypotonic-compensated intraocular pressure (IOP)

Exclusion Criteria:

* Degenerative diseases of the central nervous system, diabetes mellitus
* Primary mitochondrial dysfunction
* A history of surgical interventions and damage to the organ of vision
* Acute or chronic inflammatory or hereditary degenerative eye diseases (anterior and posterior sections)
* Decompensation of concomitant somatic diseases
* Taking antioxidants/nootropic drugs 6 months before inclusion in the study
* Hypersensitivity to ethylmethylhydroxypyridine succinate or to any of the excipients

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Degree of expression of mitochondrial dysfunction | 90 days
  Enzyme status of lymphocytes (Succinate dehydrogenase and Glycerophosphate dehydrogenase)
Dynamics of the structural and functional characteristics of mitochondria | 90 days
  Cytomorphodensitometry (number of mitochondria, their optical density, number of granules and deposits in the mitochondria of lymphocytes)

SECONDARY OUTCOMES:
Аssessment of differential light sensitivity of the retina | 90 days
  Dynamics of index of mean deviation (MD) of retinal photosensitivity [Static Automated Perimetry (SAP)]
Structural and topographic changes in the layer of nerve fibers and the retinal ganglion [Optical Coherence Tomography (OCT) parameters] | 90 days
  The average thickness of retinal nerve fibers (RNFL) of the peripapillary zone in four quadrants was studied using the Fast RNFL Thickness program and the thickness of the retinal ganglion cell complex (GCC-Ganglion Cell Complex protocol)
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 90 days
  Adverse events related to Mexidol

CONTACTS AND LOCATIONS:
Locations (1):
- Tyumen Scientific Center of the Russian Academy of Sciences, Tyumen, Russian Federation, Russia